CLINICAL TRIAL: NCT02060500
Title: Cardiaplication: A Prospective Observational Trial
Brief Title: Cardiaplication: A Novel Antireflux Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Mark L. Wulkan, M.D., Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00056015
Record Dates: First submitted 2013-12-20; First posted 2014-02-12 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; fundoplication; cardiaplication; reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiaplication (Experimental)
  Interventions: Procedure: Cardiaplication

INTERVENTIONS:
Procedure: Cardiaplication

SUMMARY:
Gastro-Esophageal Reflux is a commonly encountered problem in infants. After failure of medical therapy, many children are referred for surgical intervention. Techniques have evolved over the last 50 years; however, benefits in children remain the center of debate in many surgical forums. This is primarily owing to the high incidence of recurrence of reflux and need for revisions later in life. Some clinicians theorize that the pathophysiology of reflux in infants is different from that of the population at large, and that the traditional operation may not be the best suited for this patient population. We propose a study to test an alternative plication technique for modifying the gastro-esophageal junction at the Angle of Hiss. By plicating the cardia of the stomach, we hypothesize that we will create a valve which will limit reflux without disrupting the diaphragmatic crura, thus reducing the incidence of recurrent hiatal hernia and limiting the incidence of fundoplications which are too tight.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 12 months old who are scheduled to undergo an operative intervention for medically refractory GERD.

Exclusion Criteria:

* Inability to obtain consent
* Surgeon preference

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Determine pH impedance probe results of Cardiaplication | At 3 months post-operatively
  We will perform a pH impedance probe on all patients at 3 months post-op (+/- 30 days). We are looking for a statistically significant improvement in per-cent time the pH is <= 4.

SECONDARY OUTCOMES:
Validate elongation of the intra-abdominal esophagus as a mechanism for "outgrowing" GERD in infants | 1 year post-op
  Radiographs at 1 year will be compared to post-op chest x-ray to determine vertical length between clips placed intra-operatively at the GE junction and on the diaphragmatic crus.